CLINICAL TRIAL: NCT07372313
Title: Ability of Preoperative Carotid Artery Corrected Flow Time to Predict Hypotension and Postdural Puncture Headache During Cesarean Section
Brief Title: Prediction of Hypotension and Postdural Puncture Headache by Carotid Artery Corrected Flow Time
Status: Not yet recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Aynur Akın, professor doctor, TC Erciyes University
Other Study IDs: 2025/267
Record Dates: First submitted 2025-12-08; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Hypotension in Pregnant Women; Headache in Pregnant Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anesthesia for cesarean delivery can be provided through general or neuraxial anesthesia (spinal or epidural). Hypotension is a common complication of both methods. Hypotension associated with spinal anesthesia can cause dizziness, nausea, vomiting, restlessness, and confusion in the mother, while also decreasing blood flow to the baby, leading to hypoxia and fetal acidosis. Untreated persistent hypotension poses a life-threatening risk to both mother and baby.

In recent years, ultrasonography has become widely used to assess volume status. Carotid artery corrected flow time (FTc) is primarily affected by left ventricular preload and is related to myocardial contractility and afterload. Therefore, it can predict intraoperative hypotension.

Postdural puncture headache (PDPH) is a relatively common complication after neuraxial blocks. PDPH is generally defined as an orthostatic headache caused by low cerebrospinal fluid pressure accompanied by neck pain, tinnitus, hearing changes, photophobia, and/or nausea. Risk factors include female gender, young age, pregnancy, a previous history of PDPH, low CSF pressure, and low BMI.

This study will be conducted on pregnant women undergoing elective cesarean sections under spinal anesthesia in the cesarean operating room at Erciyes University Faculty of Medicine Hospital. The correlation between preoperative carotid artery FTc levels in pregnant women and the incidence of intraoperative hypotension and postoperative PDPH will be investigated, as will whether FTc levels are a significant predictor of the likelihood of developing intraoperative hypotension and postoperative PDPH. Carotid artery FTc will be measured 1 hour before surgery, and baseline systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), peripheral oxygen saturation (SPO2), and heart rate will be recorded in the operating room. Values will be recorded at 1, 2, 3, 5, 10, 12, 15, and 30 minutes after spinal anesthesia. Patients will be assessed postoperatively for postdural puncture headache using a numerical rating scale (NRS) on days 2, 3, and 7.

This study is expected to demonstrate the ability of preoperative FTc to predict hypotension and PDPH, to determine the threshold value for predicting hypotension and PDPH, and to improve or modify the anesthesia method in patients with predicted hypotension and PDPH.

DETAILED DESCRIPTION:
Vaginal birth is a natural and physiological process. However, in certain circumstances, a cesarean section (CS) may be necessary to protect the health of the mother and baby.

Cesarean section anesthesia can be provided through general or neuraxial anesthesia (spinal or epidural). Hypotension is a common complication in both methods.

The incidence of hypotension associated with spinal anesthesia can be as high as 74% . This condition causes dizziness, nausea, vomiting, restlessness, and confusion in the mother, while also reducing blood flow to the baby, leading to hypoxia and fetal acidosis . Hypotension lasting longer than 2 minutes is associated with a significant increase in oxypurine and lipid peroxides in the umbilical cord, indicating ischemia-reperfusion injury . Hypotension lasting less than 2 minutes does not affect neurobehavioral outcomes, while maternal hypotension lasting longer than 4 minutes can be associated with neurobehavioral changes in the first 4 to 7 days of neonatal life. Untreated persistent hypotension poses a life-threatening risk to both mother and baby.

Mechanically, spinal anesthesia-mediated sympathetic blockade affects systemic vascular resistance (SVR) and induces peripheral blood pooling, resulting in a decrease in left ventricular preload, thus causing hypotension. Aortocaval compression contributes to further preload reduction. Collateral flow decreases after spinal anesthesia, leading to severe hypotension. Therefore, monitoring techniques to assess both preload and afterload can help predict the development of hypotension and guide appropriate prophylaxis in patients.

In recent years, ultrasonography has been widely used to assess volume status. Several studies have reported that corrected blood flow time (FTc) measured in the carotid artery can predict fluid responsiveness in spontaneously breathing patients. FTc is primarily affected by left ventricular preload and is related to myocardial contractility and afterload. Therefore, it can predict intraoperative hypotension.

Accurate estimation of hypotension can improve clinical decision-making, modify anesthetic management, and facilitate early intervention.

One study reported that carotid artery FTc increased with fluid resuscitation in dehydrated patients, decreased with hemodialysis in patients with chronic kidney disease, and that the change in FTc was related to the removal of ultrafiltrate. Another study reported that pre-anesthesia carotid artery FTc in pregnant women undergoing cesarean section with spinal anesthesia may be a reliable indicator of hypotension after spinal anesthesia in women giving birth.A meta-analysis of hypotension and fluid responsiveness demonstrated that FTc exhibits superior diagnostic accuracy, particularly in the setting of anesthesia. Postdural puncture headache (PDPH) is a relatively common complication after neuraxial blocks. PDPH is a complication of dural puncture, either intentionally during spinal anesthesia or unintentionally during epidural anesthesia.

The Headache Classification Committee of the International Headache Society, in the third edition of the International Classification of Headache Disorders, defines PDPH as an orthostatic headache caused by low cerebrospinal fluid pressure, typically accompanied by neck pain, tinnitus, hearing changes, photophobia, and/or nausea. It typically occurs within five days of a lumbar puncture and is caused by cerebrospinal fluid leakage from a dural puncture. It resolves spontaneously within two weeks or after sealing the leak with an autologous epidural lumbar blood patch.

66% of PDPHs begin within the first 48 hours after a dural puncture, and approximately 90% within the first 72 hours. The typical location of the headache is frontal and occipital, radiating to the neck and shoulder region.

Risk factors include female gender, younger age, pregnancy, a previous history of PDPH, low CSF pressure, and low BMI.

Patients undergoing cesarean section carry many of the risk factors for PDPH. Therefore, predicting this would be beneficial for both the patient and the anesthesiologist.

In our literature search, we found no studies investigating the relationship between FTc and PDPH.

Carotid artery FTc offers the advantages of being noninvasive, avoiding invasive procedures, suitable for use in patients with low tidal volume or spontaneous breathing, and not affected by changes in intrathoracic pressure. As shown in many studies, it can also be used to predict hypotension. In our study, we aimed to predict intraoperative hypotension using preoperative carotid artery FTc and, unlike other studies, to investigate its relationship with postdural puncture headache.

Before starting the study, the patient and, if necessary, their relatives will be informed about the study, and their consent will be obtained. This prospective, observational study will be conducted in the cesarean operating room of Erciyes University Faculty of Medicine Hospital over a 15-month period between 2025 and 2026 on pregnant women undergoing elective cesarean sections under spinal anesthesia. The correlation between preoperative carotid FTc levels and the incidence of intraoperative hypotension and postoperative PDPH in pregnant women will be investigated, as will whether FTc levels are a significant predictor of the likelihood of developing intraoperative hypotension and postoperative PDPH.

Patients who consent to the study will fast for 6-8 hours for solid foods and 2 hours for clear liquids. One hour before surgery, they will be sent to the Doppler ultrasound room for carotid Doppler ultrasound. After a 5-minute rest in the supine position, the same radiologist will perform a Doppler ultrasound [Logiq S7/Expert (GE Healthcare; Milwaukee, WI, USA)]. The patient is supine, with their head turned 30 degrees to the left. Initially, a 6.0 to 13.0 MHz linear probe is placed vertically on the neck, with the probe pointer facing the patient's head. A long-axis B-mode image of the right common carotid artery is obtained from the inferior border of the thyroid cartilage. The probe is then placed 2 cm proximal to the carotid bifurcation, centered on the lumen. The angle between the ultrasonic beam and the blood flow direction is adjusted to less than 60 degrees. After the pulsed wave Doppler spectrum is displayed, the image is frozen. Flow time (FTc) and heart rate are measured in the carotid artery. Flow time (FTc) is measured from the beginning of the systolic upstroke to the dicrotic notch. Heart rate (HR) is obtained by measuring the interheartbeat interval at the beginning of the Doppler upstroke. FTc will be calculated using the Wodey formula after several consecutive cycles have stabilized and reached an acceptable quality level, and a single cycle will be evaluated. The Wodey formula is: FTc = FT + [1.29 × (HR - 60)]. Three separate FTc values will be calculated from three consecutive cardiac cycles, and these values will be averaged. Upon arrival to the operating room, patients will be monitored routinely, including ECG, systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), and peripheral oxygen saturation (SPO2), and baseline values will be recorded in the supine position.

As per routine practice, spinal anesthesia will be administered by an anesthesiologist not involved in the study, with the patient in a seated position, using a 26-gauge pencil-tipped spinal needle at the L3/4 or L4/5 level, and administering 0.5% hyperbaric bupivacaine according to the Hartens chart. Following the spinal injection, the patient will be placed in a supine position without any lateral tilt. Sensory block will be checked with cold and pinprick tests 3 minutes after the spinal injection and again at 6 and 9 minutes. If the sensory block level does not reach the T6 dermatome within 10 minutes, the patient will be excluded from the study.

The patient's SAB, DAB, MAP, and SpO2 will be recorded at 1, 2, 3, 5, 10, 12, 15, and 30 minutes following general anesthesia induction or spinal anesthesia administration. A 20% decrease in the patient's SAB or MAB from baseline, a decrease in SAB below 100 mmHg, or a decrease in MAP below 65 mmHg will be considered hypotension, and patients will be enrolled. As is our clinic's routine, patients with hypotension will be administered 5-10 mg ephedrine intravenously.

Patients undergoing spinal anesthesia will be evaluated for the presence of PDPH and NRS scores in person or by telephone on postoperative days 2, 3, and 7.

Statistical analysis for this study will be conducted using SPSS 22.0 (SPSS, Inc., Chicago, IL, USA).

The sample size will be determined using G-Power version 3.1.9.7 (Franz Faul, Kiel University, Germany).

Inclusion criteria were limited to patients with high cardiac risk; therefore, it was calculated that a sample of at least 84 patients would provide 95% power to detect at least a 30% difference between the 50% AUC from the null hypothesis and the 75% AUC from the alternative hypothesis.Data conformity to a normal distribution will be assessed using the Shapiro-Wilk test, and homogeneity will be assessed using the Levene test. Non-categorical data and data conforming to a normal distribution will be analyzed using a t-test between two independent groups. For data that do not conform to normal distribution and for categorical data, Chi-Square and Mann-Whitney U tests will be used to analyze the correlation between pre-anesthesia FTc and the magnitude of the decrease in SBP compared to the baseline value. Pearson correlation and/or regression analysis will be used. The area under the ROC curve will be calculated to measure the predictability of FTc in the development of hypotension. The optimal cut-off value will be determined by maximizing the Youden index. After checking for multicollinearity to measure the relationship between independent variables, a backward stepwise logistic regression analysis will be performed to evaluate the effects of age, BMI, baseline HR, SBP, DBP, and FTc on the development of hypotension. The relationship between the development of postoperative PDPH and FTc in patients undergoing spinal anesthesia will be evaluated using Pearson correlation analysis. If there is a correlation between FTc and PDPH, its direction will be determined. In all analyses, p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class II
* Regular antenatal visits
* Singleton pregnancy at ≥37 weeks' gestation
* Pregnant women aged 18-49

Exclusion Criteria:

* Patients with eclampsia or preeclampsia
* Patients who have undergone emergency cesarean section
* Patients with bleeding diatheses and those receiving anticoagulant therapy
* Patients with a history of ≥50% carotid artery stenosis
* Patients with cardiovascular disease
* Hypertension
* Patients with chronic obstructive pulmonary disease
* Patients with a heart rhythm other than sinus rhythm
* Patients with a history of cerebrovascular disease
* Patients with alcoholism or psychiatric illness
* Patients with placenta previa, accreta, or percreta
* Patients with diabetes

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women who will undergo a cesarean section with spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Predicting intraoperative hypotension using preoperative carotid artery corrected flow time (FTc). | perioperative period

SECONDARY OUTCOMES:
Post-dural puncture headache is evaluated using Numerical Rating Scales (NRS) and its relationship with preoperative corrected carotid artery flow time (FTc) is determined. | postoperative 2, 3, 7 days